CLINICAL TRIAL: NCT03783377
Title: A Phase 1 Single and Multiple Dose-Escalating Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Effects of ARO-APOC3 in Adult Healthy Volunteers as Well as in Severely Hypertriglyceridemic Patients and Patients With Familial Chylomicronemia Syndrome
Brief Title: Study of ARO-APOC3 in Healthy Volunteers, Hypertriglyceridemic Patients and Patients With Familial Chylomicronemia Syndrome (FCS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AROAPOC31001
Record Dates: First submitted 2018-12-19; First posted 2018-12-21 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Hypertriglyceridemia; Familial Chylomicronemia
MeSH Terms: conditions — Hypertriglyceridemia; Hyperlipoproteinemia Type I

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ARO-APOC3 (Experimental)
  Interventions: Drug: ARO-APOC3
- Placebo (Placebo Comparator)
  Interventions: Drug: sterile normal saline (0.9% NaCl)

INTERVENTIONS:
Drug: ARO-APOC3 — single or multiple doses of ARO-APOC3 by subcutaneous (sc) injections
  Arms: ARO-APOC3
Drug: sterile normal saline (0.9% NaCl) — calculated volume to match active treatment
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of single- and multiple doses of ARO-APOC3 in healthy adult volunteers and in patients with severe hypertriglyceridemia and familial chylomicronemia syndrome (FCS).

ELIGIBILITY:
Inclusion Criteria:

* Women of childbearing potential must have a negative pregnancy test, cannot be breastfeeding and must be willing to use contraception
* Willing to provide written informed consent and to comply with study requirements
* Normal electrocardiogram (ECG) at screening
* Hypertriglyceridemic patients must have a history of fasting serum triglycerides of at least 300 mg/dL (3.38 mmol/L) at screening or verifiable diagnosis of FCS

Exclusion Criteria:

* Clinically significant health concerns
* Regular use of alcohol within one month prior to Screening
* Use of an investigational agent or device within 30 days prior to dosing or current participation in an investigational study
* Recent use of illicit drugs
* Use of more than two tobacco/nicotine containing or cannabis products per month within 6 months prior to drug administration (applicable only to Normal Healthy Volunteers)

Note: additional inclusion/exclusion criteria may apply, per protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2021-02-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) Possibly or Probably Related to Treatment | Up to Day 113 (+/- 3 days)

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of ARO-APOC3 in Normal Healthy Volunteers (NHVs): Maximum Observed Plasma Concentration (Cmax) | Single dose phase: Up to 48 hours post-dose
PK of ARO-APOC3 in NHVs: Time to Maximum Plasma Concentration (Tmax) | Single dose phase: Up to 48 hours post-dose
PK of ARO-APOC3 in NHVs: Terminal Elimination Half-Life (t1/2) | Single dose phase: Up to 48 hours post-dose
PK of ARO-APOC3 in NHVs: Area Under the Plasma Concentration Versus Time Curve From Zero to 24 Hours (AUC0-24) | Single dose phase: Up to 48 hours post-dose
PK of ARO-APOC3 in NHVs: Area Under the Plasma Concentration Versus Time Curve From Zero to Infinity (AUCinf) | Single dose phase: Up to 48 hours post-dose
Reduction in Fasting Serum APOC3 from Pre-Dose Baseline | Up to Day 113 (+/- 3 days)

CONTACTS AND LOCATIONS:
Locations (10):
- Australia (4):
  - Research Site 2, Camperdown, New South Wales
  - Research Site 5, Sippy Downs, Queensland
  - Research Site 3, Adelaide, South Australia
  - Research Site 4, Perth, Washington
- Canada (3):
  - Research Site 7, London, Ontario
  - Research Site 6, Chicoutimi, Quebec
  - Research Site 8, Montreal, Quebec
- New Zealand (3):
  - Research Site 9, Grafton, Auckland
  - Research Site 10, Papatoetoe, Auckland
  - Research Site 11, Christchurch

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gaudet D, Clifton P, Sullivan D, Baker J, Schwabe C, Thackwray S, Scott R, Hamilton J, Given B, Melquist S, Zhou R, Chang T, San Martin J, Watts GF, Goldberg IJ, Knowles JW, Hegele RA, Ballantyne CM. RNA Interference Therapy Targeting Apolipoprotein C-III in Hypertriglyceridemia. NEJM Evid. 2023 Dec;2(12):EVIDoa2200325. doi: 10.1056/EVIDoa2200325. Epub 2023 Nov 17. PMID 38320498